CLINICAL TRIAL: NCT02719496
Title: Prove of Concept Study, to Evaluate the Efficacy, Safety, and Tolerability of IBEROGAST in the Treatment of Bowel Troubles in Patients With Parkinson's Disease
Acronym: PHYTOPARK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC15_0396
Record Dates: First submitted 2016-03-15; First posted 2016-03-25 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Gastrointestinal Disorders in Parkinson's Disease
MeSH Terms: interventions — iberogast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IBEROGAST (Experimental): Dose of 20 drops three times a day for 28 days, on constipation parkinsonian patients with disorders intestinal transit.
  Interventions: Drug: IBEROGAST

INTERVENTIONS:
Drug: IBEROGAST

SUMMARY:
The main objective of this study is to evaluate the efficacy of STW5 Iberogast, over a 28-day period, for the treatment of constipation in parkinsonian patients suffering from gastrointestinal disorders.

DETAILED DESCRIPTION:
Gastrointestinal disorders are the most common non-motor symptoms of Parkinson's disease (PD). They affect the entire intestinal tract and include excess saliva stasis (70% of patients), dysphagia (52%), gastroparesis (34-45%), and constipation. Gastroparesis participates in dyspepsia and abdominal pain. Constipation, as defined by the international standards criteria of Rome III, is present in 59% of PD patients and leads to functional impairment in 70% of patients. The mechanism underlying constipation is multifactorial and may include slow transit and defecation disorders secondary to anorectal dysfunction. Bowel disorders are present in the early stage of the disease and usually precede the onset of motor symptoms. They may result from lesions of the enteric nervous system, of the autonomic nervous system, and from probable alterations in gastrointestinal motility controlled by the central nervous system. The STW5 (Iberogast, Steigerwald, Germany) is a herbal agent composed of nine plant extracts, with prokinetic, antispasmodic, prosecretory, anti-inflammatory and anti-oxidant properties. These properties have been demonstrated in animals and in human pathology, in the treatment of dyspepsia and irritable bowel syndrome. It is the only phytotherapeutic agent which efficacy was demonstrated by randomized double-blind trials in these indications. In PD, the STW5 could improve constipation due to its prokinetic effects of the prosecretory enteric neurons. It could also improve dyspepsia and abdominal pain by its antispasmodic properties. We propose to study the efficacy and the safety of STW5 on bowel dysfunction in parkinsonian patients, especially on constipation.

ELIGIBILITY:
Inclusion Criteria:

* Patient 30 to 80 years
* Parkinson's disease according to the criteria of the United Kingdom Parkinson's Disease Society Brain Bank
* Presence of constipation defined by the Rome III criteria Functional constipation
* Social assured Patient
* Patients with signed consent

Exclusion Criteria:

* Organic Affection colic
* Constipation Drug
* Other neurological disorder Parkinson's disease
* Metabolic disease diabetes collagenoses
* Severe renal or hepatic impairment
* Pregnant or lactating women
* Premenopausal women without contraceptive device effective
* Regular and prolonged use of history (> 12 months) of laxatives irritants
* Use of oral laxative treatment in the two weeks before the start of treatment, and refusal to stop these treatment during the course of the study
* Taking treatment antabuse
* Cognitive impairment compromising understanding or application instructions
* Patient already included in a research protocol
* Minors
* Nobody protected by law

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
increasing the weekly number of exemptions of 3 in the last week of treatment compared with the reference week (Efficacity) | 28 days
  evaluate the efficacy of Iberogast, over a 28-day period, for the treatment of constipation in parkinsonian patients suffering from gastrointestinal disorders.

SECONDARY OUTCOMES:
quality of evacuations | 28 days
  weekly percentage defecation requiring thrusts, or accompanied by a sensation of incomplete rectal evacuation (agenda stool), shape and consistency of stools (Bristol scale).
Gastrointestinal Symptom Rating Scale (quality of life) | 28 days
  the impact of gastrointestinal symptoms on quality of life measured by the Gastrointestinal Symptom Rating Scale
Short Form Health Survey (SF36) (quality of life) | 28 days
  the impact of gastrointestinal symptoms on quality of life measured by the Short Form Health Survey (SF36)
use of rectal laxatives | 28 days
  use of rectal laxatives (stool diary)
clinical global improvement of gastrointestinal symptoms | 28 days
  Patient Global Impression of Change
motor and non-motor symptoms | 28 days
  Movement Disorder Society - Unified Parkinson Disease Rating Scale
Parkinson Disease Quotation ( PDQ39) (tolerability in parkinsonian) | 28 days
  Parkinson Disease Quotation ( PDQ39)
Incidence of Treatment-Emergent Adverse Events (Tolerability) | 28 days
  adverse event reporting

CONTACTS AND LOCATIONS:
Locations (1):
- Tiphaine Rouaud, Nantes, France

IPD SHARING:
Plan to Share IPD: No